CLINICAL TRIAL: NCT00682123
Title: Supplement Contamination: Detection of Nandrolone Metabolites in Urine After Administration of Small Doses of a Nandrolone Precursor
Brief Title: Risk of Positive Doping Tests Following Ingestion of Supplements Contaminated With Trace Quantities of Nandrolone Metabolites
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: UK Sport, 40 Bernard Street, London, WC1N 1ST (Unknown)
Responsible Party: Professor Ronald Maughan, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R05-P39
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Positive Doping Tests in Sports
Keywords: 19-norandrostenedione; steroids; drugs in sport; World Anti-Doping Agency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: 19-norandrostendione — Volunteers recieved 500mL of water containing 5g of creatine monohydrate and either 1.0μg, 2.5μg or 5.0μg of 19-norandrostendione in a single-blind crossover manner.
  The amount of 19-norandrostendione administered was trivial, and far less than the amounts shown to be present in many popular dietary supplements. The recommended dosage according to the distributors is 100 mg 2-3 times daily, so the administered daily dose was not more than 0.05% of the recommended dose. This dose has no measurable physiological or pharmacological effects.

SUMMARY:
There is compelling evidence that some dietary supplements consumed by the general population are manufactured and stored under conditions that lead to contamination of the end product with small amounts of extraneous materials. In most cases, this is harmless, but for athletes liable to drug testing as a consequence of their participation in sport, the potential consequences of even trivial amounts of a prohibited substance may be catastrophic. Quality control procedures for pharmaceutical products normally specify the absence of contaminants at a level of more than 0.1%, ie 1mg/g. However, in the case of an anabolic steroid such as nandrolone, the amount that will cause a positive test has been estimated to be about 1-3µg (Geyer et al, 2004). In the case of a supplement that is taken in high doses (20-30 g/d), such as for example creatine, this means that a contamination level of something closer to 0.00001% (ie 1µg/g) may cause a positive test. This work have been supported by recent findings from our laboratory (Judkins et al, 2006). These data demonstrate that as little as 10μg of 19-noradrostenedione (19-NorAD) added to a creatine supplement resulted in a positive doping test in all volunteers testing. This is one thousand times less that the purity level specified for pharmaceutical agents and at this level, these contaminants are without any pharmacological action.

Proposals are under development to regulate the sale of dietary supplements for use by athletes to avoid accidental doping positives as a result of ingestion of contaminated supplements. This requires a knowledge of the amounts of contaminant that is likely to cause problems. The aim of the present study was to examine the urinary excretion pattern of nandrolone metabolites following 1µg, 2.5µg and 5µg doses of 19-norandrostendione in both male and female subjects. The quantity of 19-norandrostenedione administered in this study is representative of the amount previously reported as an undeclared contaminant in some dietary supplements. Given the speculation surrounding positive doping cases being attributed to ingestion of sports supplements contaminated with pro-hormones, this presents an important consideration for both athletes and doping agencies, as well as supplement manufacturers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 18 - 35 years of age

Exclusion Criteria:

* Any potential participant competing in sport at a level where there is even a remote possibility of being called for a drugs test was excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Urinary 19-norandrosterone (19-NA) and 19-noretiocholanolone (19-NE) concentrations | All urine passed for 24h following supplement ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Maughan, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, School of Sport and Exercise Sciences, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Background] Geyer H, Parr MK, Mareck U, Reinhart U, Schrader Y, Schanzer W. Analysis of non-hormonal nutritional supplements for anabolic-androgenic steroids - results of an international study. Int J Sports Med. 2004 Feb;25(2):124-9. doi: 10.1055/s-2004-819955. PMID 14986195
- [Background] Maughan RJ. Contamination of dietary supplements and positive drug tests in sport. J Sports Sci. 2005 Sep;23(9):883-9. doi: 10.1080/02640410400023258. PMID 16195040
- [Background] Judkins C, Watson P, Russell C. A crossover study of 19-nor-androstenedione contamination in sports supplements: preliminary findings. Proceedings of the 5th International congress on Medical Polymers. Cologne, Germany 2006.